CLINICAL TRIAL: NCT06682546
Title: A Multicenter, Randomized, Single-blind, Etomidate-controlled, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Methoxyethyl Etomidate Hydrochloride for Sedation/Anesthesia During Gastroscopy/Colonoscopy.
Brief Title: A Trial to Evaluate the Efficacy and Safety of Methoxyethyl Etomidate Hydrochloride in Gastroscopy/Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ET-26-HCl-202
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Gastroscopy; Colonoscopy
MeSH Terms: interventions — ET-26 compound; Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ET-26 0.6 mg group (Experimental): 0.6mg/kg
  Interventions: Drug: ET-26HCl 0.6mg/kg group
- ET-26 0.8mg group (Experimental): 0.8mg/kg
  Interventions: Drug: ET-26HCl 0.8mg/kg group
- Etomidate group (Active Comparator): 0.3mg/kg
  Interventions: Drug: Etomidate Injectable Product 0.3mg/kg group

INTERVENTIONS:
Drug: ET-26HCl 0.6mg/kg group — The initial dose is 0.6 mg/kg, intravenous injection,with an additional 50% starting dose if needed (30second±5second bolus completion). Infusion time was 1minute ± 5second.
  Other Names: 0.6mg group
  Arms: ET-26 0.6 mg group
Drug: ET-26HCl 0.8mg/kg group — The initial dose is 0.8 mg/kg, intravenous injection,with an additional 50% starting dose if needed (30second±5second bolus completion). Infusion time was 1minute ± 5second.
  Other Names: 0.8mg group
  Arms: ET-26 0.8mg group
Drug: Etomidate Injectable Product 0.3mg/kg group — The initial dose is 0.3 mg/kg, intravenous injection,with an additional 50% starting dose if needed (30second±5second bolus completion).Infusion time was 1minute ± 5second.
  Other Names: 0.3mg group
  Arms: Etomidate group

SUMMARY:
A total of 78 subjects undergoing gastroscopy/colonoscopy were randomly assigned to the methoxetomidate hydrochloride group and the etomidate group according to the ratio of 1:1:1 with etomidate as the control group, 26 cases in each group. All subjects were blinded to treatment allocation. Screening assessments for all subjects will be completed within D-14 to D-2 before the first dose. For all subjects who received the investigational drug, they were required to return to the research center on D2-5 to complete the corresponding examination before being discharged from the group. To preliminarily evaluate the efficacy and safety of ET-26 in gastroscopy/colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing routine gastroscopy/colonoscopy with an expected gastroscopy/colonoscopy procedure time of less than 20 minutes;
2. age ≥ 18 and ≤ 75 years old, regardless of gender;
3. American Society of Anesthesiologists (ASA) grade I-III;
4. Body mass index (BMI) 18-30 kg/m2 (including the cut-off value) and body weight ≤100 kg;
5. Vital signs during screening: respiratory rate ≥10 and ≤24 times/min; Pulse oxygen saturation (SpO2) ≥95% while breathing air; Systolic blood pressure (SBP) ≥90mmHg and ≤160mmHg; Diastolic blood pressure (DBP) ≥60mmHg and ≤100mmHg; Heart rate (ECG) ≥55 and ≤100 beats/min;
6. Serum cortisol concentration was normal or abnormal but not clinically significant according to the investigator's judgment;
7. Able to understand the procedures and methods of this study, willing to sign the informed consent and strictly abide by the trial protocol to complete the study.

Exclusion Criteria:

1. patients requiring complex endoscopic techniques (such as cholangiopancreatography, endoscopic ultrasonography, endoscopic mucosal resection, endoscopic submucosal dissection, peroral endoscopic myotomy, etc.) or undergoing tracheal intubation;
2. patients with possible gastroduodenal outflow obstruction with retention of contents or upper gastrointestinal bleeding;
3. patients who were known or suspected to have allergies or contraindications to the components of the investigational drug or the prescribed regimen, or who were suspected to have epilepsy or severe liver and kidney dysfunction;
4. predicted difficulty in intubation or ventilation (e.g., modified Mallampti score Ⅲ-Ⅳ, congenital microglossia, mandibular hypoplasia, etc.);
5. having any of the following respiratory management risks before/at the time of screening: 1) history of asthma, wheezing; 2) sleep apnea syndrome;
6. QTcF≥450 ms (male) or ≥470 ms (female) at screening and confirmed by review; Or clinically significant electrocardiographic abnormalities that were deemed by the investigator to be ineligible for the study;
7. use of any of the following drugs or treatments before screening:1) enrolled in a clinical trial of any drug within 1 month before screening; 2) use of medications or treatments that affect cortical function within 3 days before screening; 3) Use of medications that may affect QT interval within 2 weeks before screening;
8. Laboratory tests during the screening period meet the following standards:1)AST and ALT ≥ 3×ULN;2)TBIL≥1.5×ULN;3)hemoglobin ≤90 g/L (and no blood transfusion within 14 days); 4)ANC≤1.5×109/L;5)platelet count ≤80×109/L;6)serum creatinine ≥1.5×ULN;
9. pregnant and lactating women; The reluctance of women or men of childbearing potential to use contraception for the entire dosing period; Subjects (including male subjects) who plan to become pregnant within 3 months after the trial;
10. Subjects with any other factors considered by the investigator to be ineligible for participation in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Success rate of gastroscopy/colonoscopy | within approximately 15minutes after injection
  Number of appends ≤5; No alternative medications or other sedatives/anesthetics were used from the beginning of the first dose of the trial product until the completion of gastroscopy/colonoscopy.

SECONDARY OUTCOMES:
Sedation/anesthesia success rate | Within approximately 1 minute of the end of the injection
  Percentage of subjects with a MOAA/S score ≤1 after initial dosing of the investigational drug
Duration of successful sedation/anesthesia | within approximately 1minute after injection
  The time from the first administration of the experimental drug to the MOAA/S score ≤1
Insertion duration | within approximately 7minutes after the first injection
  The time between initial administration of the investigational drug and successful insertion of the lens
Success rate of lens insertion | within approximately 7minutes after the last injection
  Percentage of subjects with successful insertion
Duration from completion of experimental drug administration to full recovery | Within approximately 30 minutes of the completion of the last injection
  The time between the completion of the last trial drug administration and the subject's full recovery (the first of three consecutive MOAA/S scores of 5)
The time from the end of treatment to full consciousness | Within approximately 30 minutes of the completion of the first injection
  The time from gastroscopy/colonoscopy withdrawal until the subject is fully awake (the first of three consecutive MOAA/S scores of 5)
Duration from the end of treatment to the end of the room | A maximum of 10 minutes after awakening
  The first occurrence time from gastroscopy/colonoscopy withdrawal to 3 consecutive departures with Aldrete score ≥9
The time when BIS reaches 60 or below | within approximately 5minutes after injection
  The period from the beginning of first dosing of the investigational product to the first BIS of 60 or less
The length of BIS between 40 and 60 | within 7minutes after injection
  Duration of BIS values between 40 and 60, including boundary values
Rate of use of remedial drugs | within 60minutes after injection
  Percentage of subjects who had used the sedative/anesthetic remedy propofol injection once or more
Test drug additions | within 30minutes after injection
  the additional situation and dosage of drugs were summarized
Cognitive function evaluation | Maximum 40 minutes after awakening
  Mini-mental State Examination

CONTACTS AND LOCATIONS:
Overall Officials: Mengchang Yang, Principal Investigator — Sichuan Academy of Medical Sciences
Locations (3):
- China (3):
  - Sichuan Academy of Medical Sciences · Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Guangyuan First People's Hospital, Guangyuan, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan

IPD SHARING:
Plan to Share IPD: No